CLINICAL TRIAL: NCT03808220
Title: Improvement in Postoperative Pain Outcome
Brief Title: Prospective Observational Study on Postoperative Pain and Side Effect
Acronym: Pain Out
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chi-Wai Cheung, Professor Cheung Chi Wai, The University of Hong Kong
Other Study IDs: UW 18-660
Record Dates: First submitted 2019-01-14; First posted 2019-01-17 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post-surgical patients: post-surgical patients > 18 years
  Interventions: Behavioral: postoperative pain intensity; Behavioral: preoperative pain frequency; Behavioral: Side effect
- pediatric patients post-op day 1: pediatric patients > 4 years on post-op day 1 (sub-project QUIPSI - PAIN OUTinfant)
  Interventions: Behavioral: postoperative pain intensity; Behavioral: preoperative pain frequency; Behavioral: Side effect

INTERVENTIONS:
Behavioral: postoperative pain intensity — estimate the postoperative pain intensity by using a scaling system via questionnaire
Behavioral: preoperative pain frequency — estimate the preoperative pain intensity by using a scaling system via questionnaire
Behavioral: Side effect — investigate the presence of any side effect

SUMMARY:
PAIN OUT is a multi-national, non-interventional registry and benchmark project, assessing and analysing clinical and patient-reported outcome data of postoperative pain.

DETAILED DESCRIPTION:
PAIN OUT offers a large registry as well as a system for benchmarking and feedback of outcome quality and decision support in acute pain conditions. It collects demographic, clinical and outcome data, using a validated assessment tool available in multiple languages.

The registry part of the project aims at performing population-based research. Furthermore, its infrastructure allows for the conduct of prospective studies comparing the effectiveness of processes of care.

The benchmark part of the project provides the medical community with a unique, user-friendly system to improve treatment of patients with postoperative pain. A web-based information system, featuring two main functions, was developed:

a feedback and benchmarking system which provides participating sites with continuously updating data and analyses about the quality of care they provide compared to other institutions and allows identification of best clinical practice.

a knowledge library which provides clinicians with easily accessible and regularly updated summaries of evidence-based recommendations tailored to specific post-operative situations.

From 2016 on, sub-projects in Mexico, China and several European countries have started. This programs take place over a period of two years during which collaborators carry out a Quality Improvement project in their hospital using methodology provided by PAIN OUT. This includes collection of baseline data in a first phase, analysis of findings according to a protocol provided by PAIN OUT, review of findings and developement of improvement measures, implementation of the improvements and assessment of outcomes after a second phase of data collection.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years or >= 4 years for sub-project QUIPSI/PAIN OUTinfant
* patient is post-op day 1
* patient is at least 6 hours on the ward
* patient has given consent

Exclusion Criteria:

* patient cannot communicate
* patient is cognitively impaired
* patient is asleep
* patient is too ill
* patient does not want to fill in the questionnaire

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adult post-surgical patients in hospitals on post-op day 1
Sampling Method: Probability Sample
Enrollment: 2197 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Questionnaire on postoperative pain treatment | first postoperative day

SECONDARY OUTCOMES:
Questionnaire on patients' perception of pain treatment outcome | first postoperative day
  questions related to worst pain since surgery, least pain since surgery, time in pain, interference of pain with activities, affect of pain on mood and emotions, pain therapy side effects, pain relief, wish for more treatment, information on treatment, participation in decisions, satisfaction, non-medical treatment methods and pre-hospital existence of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Meissner, Study Director — Jena University Hospital; Chi Wai Cheung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong